CLINICAL TRIAL: NCT06797973
Title: MOTHER Trial: Efficacy and Safety of Low-dose Intrathecal Morphine Following Planned Caesarean Section - a Randomised, Blinded, Clinical, Controlled, Multicentre Trial.
Brief Title: Efficacy and Safety of Intrathecal Morphine for Postoperative Pain Management Following Planned Caesarean Section
Acronym: MOTHER
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Anne Juul Wikkelsø (Other)
Responsible Party: Sponsor-Investigator, Anne Juul Wikkelsø, Associate Professor, Senior Consultant, PhD, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-518678-16-00; 2024-518678-16-00 (EU CTIS Number)
Record Dates: First submitted 2025-01-17; First posted 2025-01-29 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Caesarean Section; Postoperative Pain
Keywords: Caesarean section; Cesarean section; Cesarean delivery; Caesarean delivery; Postoperative pain; Intrathecal morphine; Spinal morphine; elective caesarean
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrathecal morphine (Experimental)
  Interventions: Drug: Intrathecal Morphine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo (Sodium Chloride Injection, 0.9%)

INTERVENTIONS:
Drug: Intrathecal Morphine — 80 μg preservative-free morphine (0.2 ml) added to a single-shot spinal anaesthesia consisting of 11.5 mg hyperbaric bupivacaine and 10 μg fentanyl
  Arms: Intrathecal morphine
Drug: Placebo (Sodium Chloride Injection, 0.9%) — 0.2 ml of isotonic sodium chloride added to a single-shot spinal anaesthesia consisting of 11.5 mg hyperbaric bupivacaine and 10 μg fentanyl.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if morphine added to the spinal anaesthesia can improve postoperative pain treatment for patients undergoing caesarean section, without increasing the risk of serious adverse events in mother and baby.

The main questions it aims to answer are:

* Is the treatment effective in preventing postoperative pain?
* Is the treatment safe for both mother and baby?

Participants will be given a normal spinal anaesthesia with addition of either morphine or sodium chloride (inactive substance). All participants will receive standard postoperative pain treatment, including morphine tablets as needed. Researchers will collect data from the electronic medical record and ask the participants to fill out questionnaires about pain levels and possible side effects.

DETAILED DESCRIPTION:
BACKGROUND AND OBJECTIVE:

Caesarean section is surgical procedure associated with moderate to severe postoperative pain, which can negatively affect recovery, mother-child bonding and the initiation of breastfeeding. Intrathecal morphine may offer pain relief for up to 24 hours, and is widely implemented and recommended as part of multimodal postoperative pain management. Despite the widespread use, there is limited evidence for the balance between benefits and harms of low-dose intrathecal morphine in patients undergoing caesarean section.

The objective of the trial is to evaluate analgesic efficacy as well as maternal and neonatal safety associated with addition of low-dose (80 µg) intrathecal morphine versus placebo to standard multimodal postoperative pain management in patients undergoing planned caesarean section.

The trial is a superiority, investigator-initiated, pragmatic, randomised, blinded, placebo-controlled multicentre trial.

TRIAL SIZE: A total of 1,312 participants is required to show/reject a 35% relative increase in the composite co-primary safety outcome, with an estimated baseline incidence of 21% without intrathecal morphine and a power of 80%. We adjust statistically for having two primary outcomes by using an alpha of 2.5%. We reach a power of 99.9% for the co-primary outcome of pain score with an estimated mean Numeric Rating Scale (0-10) of 4.88, standard deviation of 2.0 and relevant mean difference of 1.0.

ETHICAL CONSIDERATIONS: Intrathecal morphine for caesarean delivery represents a common medical practice which is not supported by robust evidence. High-quality data on efficacy and safety of the treatment will enable clinicians to tailor postoperative pain treatment to each patient, thus improving care for future patients. Choosing low-dose morphine minimises the risk of adverse effects, and all trial participants will receive standard multimodal pain treatment. There is no evidence of any harmful neonatal effects. All trial participants will give informed consent, and the trial will adhere to the Declaration of Helsinki as well as national and international standards of good clinical practice.

PLANNED SUBSTUDIES:

* Incidence of desaturation and bradypnea during the first 24 hours following surgery, assessed using continuous wireless respiratory monitoring in a subpopulation of 100 patients at 3 trial sites.
* Efficacy and safety of intrathecal morphine in participant subgroups: The influence of different pre-existing factors on the primary outcomes

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Singleton pregnancy
* Scheduled for planned caesarean section performed under spinal anaesthesia
* Written informed consent

Exclusion Criteria:

* Allergy to or contraindications towards trial medication
* Patients planned for postoperative epidural due to expected difficult postoperative pain management
* Patients planned for combined spinal-epidural as primary anaesthesia
* Inability to understand and read Danish
* Previous inclusion in the trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1312 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Level of pain when mobilising from supine to sitting position within 24 hours | 6, 12, 18 and 24 hours following spinal anaesthesia
  Longitudinal measurements of NRS (0-10) at 6, 12, 18 and 24 hours with most focus on the 24-hour pain level
Maternal and neonatal serious adverse events | Within 7 days from discharge
  Binary composite outcome:
  1. Death of either participant or neonate within 7 days
  2. Participants with clinically significant respiratory depression within 24 hours, defined as respiratory depression documented in the electronic medical record, e.g. need for airway management or pharmacological intervention (subjective assessment by treating clinician, validated by 2 investigators)
  3. Neonates needing admission to neonatal intensive care unit within 48 hours
  4. Hospitalisation of either participant or neonate within 7 days after discharge
  5. Participants with severe vomiting or nausea within 24 hours, defined as ≥5 points on the 'Simplified postoperative nausea and vomiting impact scale'63 at any time point (6, 12, 18 and 24 hours)

SECONDARY OUTCOMES:
Opioid consumption within 24 hours | Within 24 hours following spinal anaesthesia
  Mg oral morphine equivalents
Morphine associated adverse effects within 24 hours | Within 24 hours following spinal anaesthesia
  Binary composite outcome: participants experiencing either:
  1. Vomiting (patient reported, yes/no)
  2. Nausea
  3. Dizziness
  4. Pruritus Nausea, dizziness, and pruritus is assessed as "none", "little", "moderate", or "severe" with patients reporting "moderate" or "severe" categorised as having a positive outcome
  5. Urinary retention, defined as need for re-catheterisation within 24 hours
Obstetric quality of recovery score at 24 hours | Within 24 hours following spinal anaesthesia
  Obs-QoR-10 (0-100)
Participants satisfaction with postoperative pain-treatment during the first 24 hours | Within 24 hours following spinal anaesthesia
  NRS 0-10
Established breastfeeding at 30 days | 30 days from surgery
  Proportion of neonates being exclusively breastfed at 30 days

OTHER OUTCOMES:
Serious adverse events, pain at 24 hours and opioid consumption, compared using Win Ratio | Within 7 days from discharge
  A composite outcome analysed using Win Ratio, consisting of
  1. Maternal and neonatal serious adverse events (as defined in the primary outcome)
  2. Level of pain when mobilising from supine to sitting position at 24 hours (NRS 0-10)
  3. Opioid consumption within 24 hours (mg oral morphine equivalents)
Overall severity of pruritus within 24 hours | Within 24 hours following spinal anaesthesia
  NRS 0-10
Pharmacological treatment for opioid-related adverse effects within 24 hours | Within 24 hours following spinal anaesthesia
  Dexametasone, dosage (mg) 5-HT3 receptor antagonists, type, dosage (mg) Dopamine receptor antagonists, type, dosage (mg) Droperidol, dosage (mg) Antihistamines, type, dosage (mg) Pethidine, dosage (mg) Naloxone, dosage (mg) Clonidine, dosage (mg)
Ability to mobilise independently | 6, 12, 18 and 24 hours following spinal anaesthesia
  Proportion of participants able to mobilise independently at 6, 12, 18 and 24 hours
Level of pain at rest within 48 hours | 6, 12, 18, 24 and 48 hours following spinal anaesthesia
  Longitudinal measurements of NRS (0-10) at 6, 12, 18, 24 and 48 hours
Opioid consumption within 48 hours | Within 48 hours following spinal anaesthesia
  Mg oral morphine equivalents
"Rescue" supplemental pain treatment with truncal nerve block or epidural within 24 hours | Within 24 hours following spinal anaesthesia
  Binary composite outcome: participants receiving either an unplanned postoperative truncal nerve block or epidural analgesia within 24 hours
Level of pain when mobilising from supine to sitting position at 48 hours | Within 48 hours following spinal anaesthesia
  NRS 0-10
Total consumption of non-opioid analgesic medication (paracetamol, NSAIDs) within 24 hours and 48 hours | Within 24 and 48 hours following spinal anaesthesia
  Paracetamol, dosage (mg) NSAIDs, type, dosage (mg)
Intraoperative nausea, vomiting and pruritus | During surgery
  Binary composite outcome: participants experiencing either
  1. Intraoperative nausea
  2. Intraoperative vomiting
  3. Intraoperative pruritus Nausea and pruritus are assessed as "none", "little", "moderate", or "severe" with patients reporting "moderate" or "severe" categorised as having a positive outcome. Vomiting is assessed as yes/no.
  Intraoperative is defined as from administration of spinal anaesthesia until the patient is leaving the operating room
Overall severity of pain within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Overall severity of nausea/vomiting within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Overall severity of dizziness within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Overall severity of shivering within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Overall feeling of being comfortable within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Overall ability to mobilise independently within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Overall ability to independently hold infant within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Overall ability to nurse/feed infant independently within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Overall ability to handle personal hygiene within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Overall feeling of being in control within 24 hours (ObsQoR-10) | Within 24 hours following spinal anaesthesia
  NRS 0-10
Length of hospital stay | Within 7 days from discharge
  Total length of primary hospital stay (hours)
Readmission or unplanned hospital re-attendance within 7 days | Within 7 days following surgery
  Binary composite outcome: participants needing either:
  1. Hospital readmission within 7 days
  2. Re-attendance (unplanned hospital out-patient consultation) within 7 days
Failed or insufficient spinal anaesthesia | Within 24 hours following spinal anaesthesia
  Binary composite outcome: participants needing either:
  1. Conversion to general anaesthesia
  2. Repeated neuraxial procedure
  3. Supplemental intraoperative pain treatment
Hospital-free days within 7 days | Within 7 days following surgery
  Number of days out of hospital for both participant and neonate within 7 days
Ogilvie's syndrome/ileus within 7 days | Within 7 days following surgery
  Proportion of participants with Ogilvie's syndrome/ileus that requires surgery or treatment with neostigmine within 7 days
Apgar score at 5 minutes following birth | 5 minutes following birth
  0-10
Apgar score <7 at 5 minutes following birth | 5 minutes following birth
  Proportion of neonates with Apgar score <7 at 5 minutes following birth
Neonatal need for respiratory support within 48 hours | Within 48 hours following birth
  Proportion of neonates needing respiratory support within 48 hours, defined as either:
  1. Continuous positive airway pressure treatment
  2. Positive pressure ventilation
  3. HNF (high nasal flow)
  4. Intubation
  5. Oxygen therapy
Neonatal sedation resulting in failed breast-/bottle feeding within 48 hours | 24 and 48 hours following birth
  Proportion of neonates not being breastfed or bottle fed due to neonatal sedation, corresponding to L=0 (too sleepy or reluctant, no sustained latch or suck achieved) on the LATCH scoring system
Neonatal hospitalisation within 24 hours after discharge | 24 hours after discharge
  Proportion of neonates hospitalised within 24 hours after discharge of participant

CONTACTS AND LOCATIONS:
Locations (8):
- Denmark (8):
  - Aarhus University Hospital, Aarhus
  - Copenhagen University Hospital - Rigshospitalet, Copenhagen
  - Copenhagen University Hospital - Herlev and Gentofte, Herlev, Herlev
  - Copenhagen University Hospital - North Zealand, Hillerød, Hillerød
  - Copenhagen University Hospital - Amager and Hvidovre, Hvidovre, Hvidovre
  - University Hospital of Southern Denmark - Lillebælt Hospital, Kolding, Kolding
  - University Hospital of Southern Denmark - Odense University Hospital, Odense C
  - Zealand University Hospital, Roskilde

IPD SHARING:
Plan to Share IPD: Yes
Data supporting the findings of this study are available from the corresponding author in accordance with Danish law and upon reasonable request.